CLINICAL TRIAL: NCT03603925
Title: Enhancing SUV Accuracy of PET/MR for Clinical Trial Qualification
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE3Y18; R01CA196687 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Positron Emission Tomography-Magnetic Resonance (PET-MR)
Keywords: Computed tomography; standardized update values
MeSH Terms: interventions — Magnetic Resonance Imaging; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PET/MR + PET/CT: The interventions for participating in this research are centered around steps needed to safely and ethically collect a research PET/MR scan following a standard-of-care PET/CT scan. The patient will be imaged in at least one of several standard anatomic areas: head/neck, thorax, abdomen, pelvis or whole-body.
  Interventions: Diagnostic Test: Positron Emission Test / Magnetic Resonance (PET/MR); Diagnostic Test: Positron Emission Test / Computed Tomography (PET/CT)

INTERVENTIONS:
Diagnostic Test: Positron Emission Test / Magnetic Resonance (PET/MR) — The Philips Ingenuity PET/MR is used for research scanning. Patients receiving a clinically indicated PET/CT, will be approached to be included in this study. There is no special preparation other than that needed for the prerequisite PET/CT scanning. At the completion of the PET/CT scanning, the subject will be taken to the PET/MR scanner, which is in close in proximity, for research scanning. The research scanning would take up to one hour or as tolerated.
Diagnostic Test: Positron Emission Test / Computed Tomography (PET/CT) — Patients will receive PET / CT imaging for the detection of cancer or other clinically indicated anomalies. The completed study visit is expected to take approximately 2 hours and not longer than 3 hours.

SUMMARY:
Standardized Uptake Values (SUVs), normalized activity concentration, measured using PET/MR have inaccuracies ≥ 20% which exceeds National Cancer Institute / American College of Radiology Imaging Network (NCI/ACRIN), Radiological Society of North America / Quantitative Imaging Biomarkers Alliance (RSNA/QIBA) specifications and disqualifies PET/MR from multicenter or cooperative group clinical trials. High inaccuracy is primarily due to poor attenuation correction (AC) owing to lack of computed tomography (CT) data. This study will develop acquisition and analyses methods to synthesize CT images from MR data that can be used to achieve SUVs that are within 5% of those obtained using PET/CT (reference standard), thus meeting accuracy requirements needed to qualify for multicenter trials.

The overall goal of this research project is to validate clinically practical methods for producing MR-based attenuation correction information which is needed to produce quantitatively accurate PET images from a PET/MR scanner. Existing commercial PET/MR systems use methods that are inaccurate.

DETAILED DESCRIPTION:
Objective The primary objective is to demonstrate that, using the new acquisition and analysis methods for MR-AC, PET SUVs in lesions and normal tissues can be measured using PET/MR and be within 5% agreement of those measured using PET/CT.

The secondary objective is to demonstrate visual and quantitative agreement between synthesized CT images generated from MR data and the reference, measured CT images.

Study Design This study would like to enroll patients receiving a clinically indicated PET/CT scan. The patients will be asked to agree to a receive research PET/MR scan within the study which requires additional time and potential MR risks for the patient. It does not entail extra injections or radiation exposure. Research acquisition and processing will be performed on the PET/MR data to create PET images that are expected to have quantitatively accurate SUVs. These will be compared to SUVs from the clinical PET/CT which will serve as the reference standard.

Outcome By bringing together cutting-edge advances in both MR acquisition and image analyses, the successful completion of these aims will achieve SUVs that are within 5% of those obtained with PET/CT (reference standard) with clinically appropriate acquisition time, image quality, and diagnostic accuracy, so that PET/MR systems meet SUV accuracy requirements needed to qualify for cooperative group clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Receiving PET/CT at University Hospitals Cleveland Medical Center (UHCMC) for a clinical indication
* No Contraindications to undergo MR as assessed using University Hospitals (UH) Radiology standard MR assessment form
* Has the ability to understand and willingness to sign a written informed consent
* The circumference of the volunteer in the body section, as determined using a measuring tape, to be scanned must be less than or equal to 110 cm to avoid field of view limitations on the PET/MR

Exclusion Criteria:

* Patient size or circumference greater than the MR gantry of the PET/MR.
* Pregnancy or lactation.
* Contraindications to undergo MR as assessed using UH Radiology standard MR assessment form.
* Claustrophobia or inability to tolerate MR examination (lay still for approximately 1 hour and hold breath intermittently).
* Individuals who are not willing or capable of giving informed consent or assent (with legal guardian consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving PET/CT at University Hospitals Cleveland Medical Center (UHCMC) for a clinical indication
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Quantitative agreement between measured CT and CT synthesized from MR data (Hounsfield Units) | Up to 3 hours after beginning scan
  Demonstrate quantitative agreement between measured CT and CT synthesized from MR data
Quantitative agreement in the derived linear attenuation coefficients at 511 kilo electro volts (keV). | Up to 3 hours after beginning scan
  Demonstrate quantitative agreement in the derived linear attenuation coefficients at 511 keV.

SECONDARY OUTCOMES:
Percent difference in Standardized Uptake Values (SUVs) in PET/CT scans compared to PET/MR scans | Up to 3 hours after beginning scan
  Demonstrate that SUVs in lesions and normal tissues measured using MR-based attenuation correction (MR-AC) are within 5% of those measured using PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F. Muzic, PhD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States